CLINICAL TRIAL: NCT04876287
Title: Salivary dysfuncTion After Radioiodine Treatment
Acronym: START
Status: Completed | Type: Observational
Sponsor: Institut de Radioprotection et de Surete Nucleaire (Other Government)
Responsible Party: Principal Investigator, Clemence BAUDIN, Principal Investigator, Institut de Radioprotection et de Surete Nucleaire
Other Study IDs: 2020-A00208-31
Record Dates: First submitted 2021-04-26; First posted 2021-05-06 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Thyroid Cancer
Keywords: radioiodine; salivary dysfunctions; genetic polymorphism; dosimetry
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Iodine-131

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients treated by 1.1 GBq
  Interventions: Drug: Radioiodine
- patients treated by 3.7 GBq
  Interventions: Drug: Radioiodine

INTERVENTIONS:
Drug: Radioiodine — cancer therapy

SUMMARY:
Aim/Introduction:

The treatment of differentiated thyroid cancer includes generally a total thyroidectomy, followed by a radioiodine (131I)-therapy. Due to their ability to concentrate iodine, the salivary glands may present inflammation after administration of 131I, which may be symptomatic, may lead to longer-term chronic abnormalities, resulting in alterations in patients' nutrition and quality of life. The incidence of salivary dysfunctions after 131I-therapy varies considerably between studies due to methodological limitations. Also, the occurrence of these dysfunctions may be linked to increased uptake and/or retention of 131I in the salivary glands and/or individual radiosensitivity. However, no clinical or genetic factors have been identified to date to define patients at risk, allowing the delivered activity to be adapted to the expected risk of salivary dysfunctions. The aims of this study are to estimate the incidence of salivary dysfunctions after 131I-therapy, to characterize patients at risk of developing post-treatment dysfunctions using clinical, biomolecular and biochemical factors, and to validate a dosimetric method to calculate the dose received at the salivary gland level in order to analyse the dose response relationship between exposure of salivary glands to 131I and salivary dysfunctions.

Materials and Methods:

This prospective cohort aims to include 120 patients, candidates for a 131I-therapy in the context of their differentiated thyroid cancer, treated in the Nuclear Medicine department of the Pitié-Salpêtrière hospital (40 and 80 patients in a 1.1GBq and a 3.7GBq dose groups respectively). The follow-up is based on 3 scheduled visits: at inclusion (immediately before 131I therapy), 6months and 18months after treatment. For each visit, questionnaires on salivary disorders (validated French tool), quality of life (HAD-scale, MOS-SF-36), and nutritional status are administered. At inclusion and at T6, saliva samples and individual measurement of the salivary flow, without and with salivary glands stimulation, are performed.

External thermoluminescent dosimeters are placed opposite the salivary glands and at the sternal fork on the treatment's day before radioiodine administration and removed 5days after treatment. From dosimeters, a reconstitution of the dose received at the salivary glands will be established using physical and computational phantoms.

Genetic and epigenetic analyses will be performed to find biomarkers of predisposition to develop salivary disorders after 131I-therapy.

Expected results Inclusion of patients started in September 2020 and are still ongoing. Statistical analyses will study the links between salivary dysfunctions and the 131I dose received by the salivary glands, taking into account associated factors. In addition, impacts on the patients' quality of life will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* treated for differencied thyroid cancer
* aged of 18 and more

Exclusion Criteria:

* having been treated by chemiotherapy or radiotherapy
* no French language
* can't be follow at 6 months after treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
decrease in salivary flow (mL) after radioiodine therapy | 6 months
  salivary flows (with and without stimulation of the salivary glands) are measured before and 6 months after the radioiodine treatment. A decrease of 5% of the flows will allow to caracterize the outcome 1
Anxiety and depression symptoms | 18 months
  The Hospital Anxiety and Depression (HAD) validated scale will be use to assess the outcome 2.
  The HAD scale is an instrument that screens for anxiety and depressive disorders. It includes 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus making it possible to obtain two scores (maximum score for each score = 21).
  To screen for anxiety and depressive symptomatology, the following interpretation will be adopted for each of the scores (A and D):
  * 7 or less: no symptomatology
  * 8 to 10: doubtful symptomatology
  * 11 and more: definite symptomatology.
Eyes dryness | 18 months
  The Ocular Surface Disease Index (OSDI) will be use for eye dryness assessment. It is assessed on a scale of 0 to 100, with higher scores representing greater disability.
  The index demonstrates sensitivity and specificity in distinguishing between normal subjects and patients with dry eye disease. The OSDI© is a valid and reliable instrument for measuring dry eye disease severity (normal, mild to moderate, and severe) and effect on vision-related function.
Self-rating Quality of life | 18 months
  The Medical Outcomes Study (MOS) 36-item short-form (SF-36) includes one multi-item scale that assesses eight health concepts: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions.
  The arithmetic averaging of the SF-36 domains scores will be used. For each domain, a score will be calculated from 0 to 100, with a greater score indicating a better-perceived health state. These 8 scales wil be compressed into 2 primary summary scales: The physical component scale (PCS) and the mental component scale (MCS). An overall (global) SF-36 score was calculated by summating the 8 dimensions and dividing by 8.
Salivary dysfunctions | 18 months
  A French validated questionnaire (no name) fomr Moreddu at el. (2017) will be used to assess salivary dyfunctions. The questions concerned discomfort, pain, hyposialorrhoea, and quality of life. Nine of the 13 questions use nominal variables (Yes/No), and two use ordinal variables. A visual analogue scale (VAS) is also included into the questionnaire to evaluate the intensity of pain (greater score for higher pain, from 0 to 10). The outcome 5 will be determined with at least 1 "yes" to a nominal question or a score >7 at the VAS.
Nutrition | 18 months
  The EVA (échelle visuelle analogique) will be used to asses a decrease in nutrition with a score between 0 and 10. A score less than 8 will determine troubles in nutrition.

CONTACTS AND LOCATIONS:
Locations (1):
- Pitié-Salpêtrière hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baudin C, Bressand A, Buffet C, Menegaux F, Soret M, Le AT, Cardon T, Broggio D, Bassinet C, Huet C, Armengol G, Richardson DB, Leenhardt L, Bernier MO, Lussey-Lepoutre C. Dysfunction of the Salivary and Lacrimal Glands After Radioiodine Therapy for Thyroid Cancer: Results of the START Study After 6-Months of Follow-Up. Thyroid. 2023 Sep;33(9):1100-1109. doi: 10.1089/thy.2023.0090. Epub 2023 Jun 23. PMID 37300484
- [Derived] Baudin C, Lussey-Lepoutre C, Bressand A, Buffet C, Menegaux F, Soret M, Broggio D, Bassinet C, Huet C, Armengol G, Leenhardt L, Bernier MO. Salivary Dysfunctions and Consequences After Radioiodine Treatment for Thyroid Cancer: Protocol for a Self-Controlled Study (START Study). JMIR Res Protoc. 2022 Jul 22;11(7):e35565. doi: 10.2196/35565. PMID 35867385